CLINICAL TRIAL: NCT04288830
Title: Evaluation of a Tai Chi Resilience Training Program on Objective and Subjective Measures of Post Traumatic Stress Disorder Severity
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: IRB00226155
Record Dates: First submitted 2020-02-26; First posted 2020-02-28 (Actual); Last update posted 2023-04-11 (Actual); Status verified 2023-01

CONDITIONS: Post Traumatic Stress Disorder; Tai Chi; Aerobic Exercise
MeSH Terms: conditions — Stress Disorders, Post-Traumatic | interventions — Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- TCMMMRT First (Experimental): Participants will perform an instructor-led mind-body exercise regimen 1 day per week during this arm of the study for a total of 8 weeks. Home practice will be logged. At the completion of the TCMMMRT Condition, participants will perform an instructor-led low impact aerobic exercise regimen 1 day per week for a total of 8 weeks. Home exercise will be logged.
  Interventions: Behavioral: Tai Chi Moving Mindfulness Meditation and Resilience Training; Behavioral: Aerobic Exercise
- Aerobic Exercise First (Active Comparator): Participants will perform an instructor-led low impact aerobic exercise regimen 1 day per week during this arm of the study for a total of 8 weeks. Home exercise will be logged. At the completion of the aerobic exercise condition, participants will perform an instructor-led mind-body exercise regimen 1 day per week for a total of 8 weeks. Home practice will be logged.
  Interventions: Behavioral: Tai Chi Moving Mindfulness Meditation and Resilience Training; Behavioral: Aerobic Exercise

INTERVENTIONS:
Behavioral: Tai Chi Moving Mindfulness Meditation and Resilience Training — Low-impact mind-body exercise adapted from traditional tai chi.
Behavioral: Aerobic Exercise — Low-impact aerobic exercise, led by instructor

SUMMARY:
The standard of care for PTSD involves both psychotherapy and pharmacotherapy, but treatment resistance is common. The discovery of effective complementary treatment approaches would have major implications for patients with PTSD. Mindfulness meditation and related practices have been studied intensively in recent years for a variety of psychiatric illnesses, including depression, generalized anxiety disorder, and PTSD. Studies in PTSD suggest that mindful meditation holds promise. For example, mindfulness-based stress reduction (MBSR) has shown effectiveness for reducing symptom severity and improving mental-health related quality of life in combat-exposed veterans and child survivors of sexual abuse. Mechanistically, mindfulness meditation appears to counteract the types of functional changes that have been identified in the brains of patients with PTSD. In particular, while PTSD symptoms are associated with decreased activation of the prefrontal cortex (PFC) and increased amygdala activity, mindfulness meditation is associated with increased PFC activation and decreased amygdala activation. Other physiological effects of mindfulness meditation in patients with PTSD are not fully defined. However, available data suggest that it leads to a normalization of vagal tone and plasma cortisol levels, which are known to be abnormal in patients with chronic PTSD. Research utilizing validated and standardized pre- and post- PTSD outcome measures, in addition to pre- and post- physiologic variables such a vagal tone, plasma cortisol and catecholamine levels, may better the understandings of physiological effects of mindfulness medication.

DETAILED DESCRIPTION:
Post-traumatic stress disorder (PTSD) affects an estimated 4.7% of the United States population every year, leading to increased rates of disability, suicide, substance use, and interpersonal difficulties. Mindfulness interventions for PTSD offer a low-cost, repeatable method that has the potential to induce fear extinction, and that has no known side effects. While several studies have reported the efficacy of mindfulness meditation and related mind-body exercises to reduce self-reported PTSD symptoms, little is known about the physiologic changes associated with mindfulness interventions. The present study seeks to evaluate the effects of a mind-body mindfulness intervention (tai chi) on subjective reports of PTSD symptoms, as well as physiologic correlates of PTSD in a population of law enforcement officers. Tai chi was chosen because its focus on awareness of physical movements is expected to provide an easier mindfulness target, as compared to traditional seated meditation. It is well documented that patients with PTSD, who frequently struggle with intrusive trauma-related memories, are often unable to attend to current circumstances, a problem that leads to exacerbation of symptoms. While there are promising preliminary data suggesting that tai chi leads to improvements in self-reported symptoms of PTSD, there are no data regarding the effects of tai chi on objective endocrine, physiological, and behavioral measures of PTSD.

The investigators hypothesize that the use of the mind-body practice of tai chi will lead to reductions in subjective self-report measures of PTSD as well a normalization of objective physiological correlates of PTSD. In particular, it is hypothesized that the efficacy of tai chi in the treatment of PTSD is hypothesized to be achieved by facilitating fear extinction and augmenting stress resilience through improved integration of mindfulness practices with daily physical activities. To test this hypothesis, the investigators propose the following specific aims:

• Specific Aim 1: To determine the self-reported symptom changes, behavioral changes, and physiological effects that take place during an 8-week intervention of simplified Tai Chi Moving Mindfulness Meditation and Resilience Training (TCMMMRT) in a population of police officers with and without self-reported PTSD. Results from these two groups will also be compared to a control group engaging in aerobic exercise.

* Self-reported outcome measures: Brief Pain Inventory (BPI) short form, Beck Depression Inventory (BDI), Pittsburgh Sleep Quality Index (PSQI), PTSD Checklist for Diagnostic and Statistical Manual of Mental Disorders (DSM-V) (PCL-5), and Canadian Occupational Performance Measure (COPM).
* Physiological outcome measures: Mobile Acoustic startle Reflex-monitoring System (MARS) measures, heart rate variability (HRV), cortisol measurements, and actigraphy to monitor sleep patterns and activity levels.

ELIGIBILITY:
Inclusion Criteria:

For inclusion as a healthy control or a participant with PTSD:

* working in law enforcement
* between the ages of 18 and 65
* Both men and women

For inclusion as a participant with PTSD:

* previously diagnosed with PTSD by a medical professional (For inclusion in the PTSD group)
* Must meet criteria for PTSD as determined by the PCL-5 instrument on the day of initial assessment.

Exclusion criteria:

* taking sedative or stimulant drugs daily
* physical illness, injury, or disability preventing safe execution of low impact aerobic exercise

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 63 (Actual)
Dates: Start 2021-10-15 (Actual); Primary Completion 2022-07-27 (Actual); Study Completion 2022-07-27 (Actual)

PRIMARY OUTCOMES:
Change in PCL-5 Score | Assessed on Day 1, Day 56, Day 112, and Day 168
  Score on the PTSD Symptom Checklist for DSM-5. The PTSD Checklist for DSM-5 (PCL-5) is a 20-item self-report measure that assesses the presence and severity of PTSD symptoms. Items on the PCL-5 correspond with DSM-5 criteria for PTSD. The PCL-5 can be used to quantify and monitor symptoms over time, to screen individuals for PTSD, and to assist in making a provisional or temporary diagnosis of PTSD.

SECONDARY OUTCOMES:
Change in BPI score | Assessed on Day 1, Day 56, Day 112, and Day 168
  Brief Pain Inventory - a 9 item self-administered questionnaire used to assess pain severity and the affect of pain on daily functioning. Contains four measures of pain severity on a 0-10 scale and pain interference with 7 life activities on a 0-10 scale. It also includes items to specify pain location and treatments attempted. Across all numbered scales, higher numbers indicate more pain.
Change in BDI score | Assessed on Day 1, Day 56, Day 112, and Day 168
  Beck Depression Inventory - a 21 item assessment of depressive symptoms. Raw score of 0-13 indicates minimal depression, 14 to 19 indicates mild depression, 20-28 indicates moderate depression, 29-63 indicates severe depression.
Change in PSQI score | Assessed on Day 1, Day 56, Day 112, and Day 168
  Pittsburgh Sleep Quality Index - a 19 item assessment of different aspects of sleep that yields seven component scores and one component score. The composite scores range from 0 to 21, where lower scores denote a healthier sleep quality. Components are subjective sleep quality, sleep latency, sleep duration, habitual sleep efficiency, sleep disturbances, use of sleeping medication, and daytime dysfunction.
Change in COPM score | Assessed on Day 1, Day 56, Day 112, and Day 168
  Canadian Occupational Performance Measure - a semi-structured interview that enables assessment of occupational performance problems. It results in two scores of participant-perceived levels of occupational performance. It results in two main scores, performance and satisfaction, each out of 10, with higher numbers reflecting greater performance and satisfaction.
Change in Salivary Cortisol | Assessed on Day 1, Day 56, Day 112, and Day 168
  Cortisol level in mcg/dL obtained from saliva sample.
Change in Heart Rate Variability | Assessed on Days 1, 7, 14, 21, 28, 35, 42, 49, 56, 63, 70, 77, 84, 91, 98, 105, 112, and Day 168
  Heart Rate Variability collected using non-invasive Actigraph. Beat to beat intervals will be recorded by the device and output as the standard deviation of nearest neighbor (SDNN) and the square root of the means of the squares of the successive differences between adjacent nearest neighbors (RMSSD).
Change in Acoustic Blink Response | Assessed on Days 1, 7, 14, 21, 28, 35, 42, 49, 56, 63, 70, 77, 84, 91, 98, 105, 112, and Day 168
  Response to an acoustic tone (milliseconds from tone to eye blink) collected using the Mobile Acoustic startle Reflex-monitoring System (MARS) device

CONTACTS AND LOCATIONS:
Overall Officials: Una McCann, Principal Investigator — Johns Hopkins University
Locations (1):
- Johns Hopkins Bayview Medical Center, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No